CLINICAL TRIAL: NCT04576338
Title: "Neighborhood Disadvantage, Sleep, and Vascular Health: Racial Disparities in Cardiometabolic Health and Blood Pressure"
Brief Title: "Neighborhood Disadvantage, Sleep and Vascular Health"
Acronym: NDSVH
Status: Completed | Type: Observational
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Austin Robinson, Assistant Professor, Auburn University
Other Study IDs: AU IRB #20-262 FB
Record Dates: First submitted 2020-09-19; First posted 2020-10-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure; Sleep; Racism; Stiffness, Arterial; Endothelial Dysfunction
Keywords: blood pressure; sleep; endothelial dysfunction; social determinants of health; arterial stiffness
MeSH Terms: conditions — Racism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The investigators will store plasma, serum, and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- College Students: The cohort consists of Black and White college students at a university in a southeastern state in America.

SUMMARY:
The purpose of the study is to find out the effects of neighborhood disadvantage and sleep disparities contribute to racial disparities in cardiometabolic health and blood pressure in young adults.

DETAILED DESCRIPTION:
There are well-documented disparities between Black and white Americans in the incidence of cardiovascular disease, the leading cause of death in America. There are also disparities between Black and White Americans in the incidence of hypertension (high blood pressure; BP), which is the leading risk factor for cardiovascular disease. Our long-term goal is to determine effective strategies to prevent racial disparities in cardiovascular health. In this proposal, the investigators will focus on determining societal and biological mediators of racial disparities in young adults that can be targeted in future interventions. Poor sleep is associated with adverse cardiovascular events and hypertension. Moreover, recent meta-analyses demonstrate that Black adults have consistently poorer sleep health than White adults, including receiving fewer total sleep minutes and having worse overall sleep quality. Neighborhood socioeconomic environments influence health behaviors through both material resources (e.g., access to healthful foods and safe public space) and social norms (e.g. exercise, diet, smoking). A well-documented history of discriminatory policies and practices has resulted in black individuals living in more disadvantaged physical and social environments than whites. As such, they experience greater adverse exposures (e.g., racism, violence and stress), which negatively impact sleep, resulting in dysregulation of cardiometabolic health. Therefore, the investigators seek to determine the role of neighborhood disadvantage and sleep in contributing to racial disparities in cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Systolic blood pressure greater than 150 mmHg
* Diastolic blood pressure greater than 90 mmHg
* Body mass index above 35 kg/m^2
* History of cardiovascular disease
* Recent (one year) history of cancer
* History of metabolic disease (e.g. type 2 diabetes)

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The cohort consists of Black and White college students at a university in a southeastern state in America. The cohort will be, by design, generally healthy, young adults free from known cardiometabolic disease,
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) | Baseline racial comparison
  Flow-mediated vasodilation will be assessed using continuous measures of brachial artery diameter and velocity via duplex Doppler ultrasound (Hitachi Arietta 70). The brachial artery will be imaged in the longitudinal plane proximal to the medial epicondyle using a high-frequency (6-12 MHz) linear-array probe. The ultrasound probe will be stabilized using a custom-built clamp. Shear rate (sec-1) will be calculated as [(blood flow velocity (cm*s-1) *4)/blood vessel diameter (mm)] The image will be recorded throughout a 60-s baseline, a 300-s ischemic stimulus (250 mmHg), and 180 seconds post deflation. FMD will be expressed as % dilation (final diameter-baseline diameter/baseline diameter x 100) and also normalized to the shear stimulus. Allometric scaling will be used if appropriate, including if there are baseline differences in artery diameter by race or condition.
Pulse wave velocity (arterial stiffness) | Baseline racial comparison
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV). A high-fidelity strain-gauge transducer is used to obtain the pressure waveform at the carotid pulse. Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded.PWV will be expressed as cm/s.
Pulse wave analysis (arterial stiffness) | Baseline racial comparison
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) using an upper arm blood pressure cuff. PWA will be expressed as % (calculated as augmentation pressure divided by the pulse pressure).
24-hour ambulatory blood pressure | Baseline racial comparison
  Participants will wear an Oscar2 (with SphygmoCor) ambulatory blood pressure monitor on their upper arm for up to 24-hours preceding their study visit to measure systolic and diastolic blood pressure. The purpose of the ambulatory blood pressure monitoring is to determine blood pressure regulation over an entire day. This blood pressure monitor will be set to automatically take blood pressure every 20 minutes. The monitor records and saves each blood pressure measurement automatically.
Blood pressure reactivity | Baseline racial comparison
  The investigators will measure systolic and diastolic pressure using photoplethysmography at the finger. Systolic and diastolic blood pressure will be assessed at rest and during handgrip exercise. Blood pressure reactivity will be expressed as a change in pressure (mmHg) from baseline to a predetermined time during the stressor (e.g., minute one average and minute two average).
Objective sleep duration and quality | Baseline racial comparison
  Philips actiwatch spectrum will be used to quantify sleep duration. Participants will wear the watch units for 7 days. The investigators will cross-check actigraphy wear times with a sleep diary.
Subjective sleep quality | Baseline racial comparison
  The investigators will use the Pittsburgh Sleep Quality Index (PSQI) to asses sleep duration and perceived sleep quality reflective of the one month period leading into the study. The PSQI global score has a possible range of 0-21 points.

SECONDARY OUTCOMES:
Circulating reactive oxygen species | Baseline racial comparison
  The investigators will use electron paramagnetic resonance to measure reactive oxygen species (spectra units) in whole blood samples treated with a spin probe.
Blood biomarkers of nitric oxide bioavailability | Baseline racial comparison
  The investigators will measure nitric oxide metabolites (nitrate and nitrite nanomolar concentration) using chemiluminescence
Physical activity | Baseline racial comparison
  Participants will wear an ActiGraph GT3X accelerometer for seven days to objectively quantify steps per day and metabolic equivalents per day.
Mental health - social anxiety | Baseline racial comparison
  The investigators will administer the Liebowitz Social Anxiety Scale. The scale starts at 0 (none) and ends at 3 (severe) for 24 questions related to anxiety and avoidance, and a cumulative score is calculated.
Mental health - depression | Baseline racial comparison
  The investigators will administer the Beck's Depression Inventory. The scale starts at 0 and ends at 3 for 21 questions related to depression.
Neighborhood disadvantage | Baseline racial comparison
  The investigators will ask participants to identify their home addresses with investigator assistance and Google maps and potential assistance from their guardians or parents during early- and mid-childhood and adolescence. The investigators will use the participant's address and census tract information to determine measures of neighborhood quality such as median income, crime rates, and median education level.
Habitual dietary intake | Baseline racial comparison
  The investigators will instruct participants to complete a diet log for 5 days which will be operationalized with Nutrition Data System for Research (NDSR).

OTHER OUTCOMES:
24-hour urine electrolytes | Baseline racial comparison
  The investigators will use an electrolyte analyzer to assess sodium, potassium, and chloride concentration. The investigators will use urine volume and electrolyte concentration to determine 24-hour electrolyte excretion

CONTACTS AND LOCATIONS:
Overall Officials: Austin T Robinson, PhD, Principal Investigator — Auburn University
Locations (1):
- Kinesiology Building, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate DMDA approvals
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following study completion, indefinitely
Access Criteria: Upon reasonable request such as request to collaborate, performing a meta-analysis, or determine reliability, data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate DMDA approvals.

REFERENCES:
- [Result] Jeong S, Linder BA, Barnett AM, Tharpe MA, Hutchison ZJ, Culver MN, Sanchez SO, Nichols OI, Grosicki GJ, Bunsawat K, Nasci VL, Gohar EY, Fuller-Rowell TE, Robinson AT. Interplay of race and neighborhood deprivation on resting and ambulatory blood pressure in young adults. Am J Physiol Heart Circ Physiol. 2024 Sep 1;327(3):H601-H613. doi: 10.1152/ajpheart.00726.2023. Epub 2024 Jul 12. PMID 38995211
- [Result] Robinson AT, Linder BA, Barnett AM, Jeong S, Sanchez SO, Nichols OI, McIntosh MC, Hutchison ZJ, Tharpe MA, Watso JC, Gutierrez OM, Fuller-Rowell TE. Cross-sectional analysis of racial differences in hydration and neighborhood deprivation in young adults. Am J Clin Nutr. 2023 Oct;118(4):822-833. doi: 10.1016/j.ajcnut.2023.08.005. Epub 2023 Aug 22. PMID 37619651
- [Derived] Culver MN, Linder BA, Lyons DE, Hutchison ZJ, Garrett CL, McNeil JN, Robinson AT. Do not sleep on vitamin D: vitamin D is associated with sleep variability in apparently healthy adults. Am J Physiol Regul Integr Comp Physiol. 2025 Mar 1;328(3):R262-R273. doi: 10.1152/ajpregu.00168.2024. Epub 2025 Jan 28. PMID 39873709
- [Derived] Jeong S, Linder BA, Barnett AM, Tharpe MA, Hutchison ZJ, Culver MN, Sanchez SO, Nichols OI, Grosicki GJ, Bunsawat K, Nasci VL, Gohar EY, Fuller-Rowell TE, Robinson AT. Interplay of Race and Neighborhood Deprivation on Ambulatory Blood Pressure in Young Adults. medRxiv [Preprint]. 2023 Sep 12:2023.09.11.23295160. doi: 10.1101/2023.09.11.23295160. PMID 37745604